CLINICAL TRIAL: NCT01161095
Title: A Multicenter Analysis of Levonorgestrel-Intrauterine System (LNG-IUS) Use in the Postpartum Period
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No recruitment occurred and the PI stopped the study.
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCP.2010.0074
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Contraception; Postpartum Period
Keywords: Intrauterine Device; Postpartum contraception; Long-acting reversible contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate (Experimental): LNG-IUS insertion within the timeframe of delivery of the placenta to 72 hours postpartum
  Interventions: Device: LNG-IUS
- Interval (Active Comparator): LNG-IUS insertion after 6 weeks postpartum
  Interventions: Device: LNG-IUS

INTERVENTIONS:
Device: LNG-IUS — Mirena (Bayer)- Levonorgestrel-Intrauterine System

SUMMARY:
The primary objective of the investigators study is to determine if there is a difference in continuation rates at six months in women who are randomized to have the Levonorgestrel Intrauterine System (LNG-IUS) inserted at two possible time periods: Immediate (defined as after delivery of placenta to 72 hours postpartum) or Interval (defined as after 6 weeks postpartum).

DETAILED DESCRIPTION:
The control arm of our study will be women who are randomized to receive LNG-IUS in the Interval time period. The study arm will consist of women randomized to receiving Immediate placement.

The investigators hypothesize that Immediate placement of IUD in the postpartum period will result in a 20% decrease in continuation rates at six months compared to Interval placement.

Secondary outcome measures that we will obtain include:

* Pain at the time of placement
* Postpartum Depression
* Breastfeeding status
* Postpartum weight retention
* Expulsion Rates
* Bleeding Profile
* Uterine Infection(Endometritis)

ELIGIBILITY:
Inclusion Criteria:

* All women >37 weeks gestation who desire LNG-IUS for postpartum contraception who do not have a contraindication as described below will be offered participation in our study.

Exclusion Criteria:

Contraindications to the LNG-IUS include:

* Pregnancy or suspicion of pregnancy
* Congenital or acquired uterine anomaly including fibroids if they distort the uterine cavity
* Postpartum endometritis within the past 3 months
* Known or suspected uterine or cervical neoplasia or unresolved, abnormal pap smear
* untreated acute cervicitis or vaginitis including bacterial vaginosis or other lower genital tract infections
* acute liver disease or liver tumor
* hypersensitivity to any component of the product
* known or suspected carcinoma of the breast

Any of these conditions would exclude the patient from receiving these forms of contraception in our study.

In addition the following intrapartum findings, the following would exclude the patient:

* Delivery <37 weeks
* Intrapartum chorioamnionitis (defined as maternal fever >100.4 and two of the following conditions: Maternal leukocytosis (greater than 15,000 cells/cubic millimeter), Maternal tachycardia (greater than 100 beats/minute), Fetal tachycardia (greater than 160 beats/minute), Uterine tenderness, Foul odor of the amniotic fluid
* Postpartum Hemorrhage (defined as >500cc EBL for spontaneous vaginal delivery or >1000cc for cesarean delivery)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2014-05-28 (Actual); Study Completion 2014-05-28 (Actual)

PRIMARY OUTCOMES:
Continuation Rates | 6 months
  Primary objective: Determine if there is a difference in continuation rates at six months postpartum in women who have the Levonorgestrel Intrauterine System (LNG-IUS) inserted at two time periods: Immediate (after delivery of placenta to 72 hours postpartum) or Interval (after 6 weeks postpartum).
  Our analysis will be conducted on all randomized women on an intention to treat basis. Once insertion has occurred, evaluation at 6 months postpartum with the presence or absence of the LNG-IUS in the uterus will be determined to calculate the continuation rate.

SECONDARY OUTCOMES:
Pain at insertion | 1 minute
  Pain will be measured using the validated Visual Analog Scale (VAS) at the time of insertion.
Postpartum Depression | 6 months
  Depression history will be determined from the initial data collection sheet upon entry into the study. The Edinburgh Postnatal Depression Scale will be filled out by the participant at their six week postpartum appointment (routine), and also at six months.
Breastfeeding Status | 6 months
  We will identify those who plan on breastfeeding their infants prior to discharge from the hospital. We will also determine the number of hours to Lactogenesis II (avg 40-50 hrs) via phone interview within one week from discharge. We will determine discontinuation rates and days to discontinuation of breastfeeding at six weeks and six months. We will also record infant weights at the postpartum appointment and at six months.
Postpartum weight retention | 6 months
  We will determine each participant's pre pregnancy BMI, BMI at admission to labor and delivery, and BMI at the postpartum appointment and at 6 months.
Sexual Function | 6 months
  We will determine the number of days from delivery to resumption of sexual intercourse. We will also have the participant complete the Female Sexual Function Index questionnaire (FSFI) at the postpartum appointment and at 6 months.
Expulsion Rate | 6 months
  Expulsion rate as well as resumption of contraception (whether LNG-IUS is replaced or another form of contraception is initiated) occurs at the postpartum appointment and at six months
Bleeding Profile | 6 months
  Each Participant will be asked to complete a monthly menstrual flow calendar to document light, medium, or heavy bleeding. These will be collected at the postpartum appointment and at six months.
Infectious morbidity | 6 months
  Postpartum endometritis and pelvic inflammatory disease will be tracked with record review and direct participant questioning at their postpartum appointment and at six months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Arkansas for the Medical Sciences, Little Rock, Arkansas
  - Naval Medical Center, Portsmouth, Virginia